CLINICAL TRIAL: NCT00000890
Title: Effect of Highly Active Antiretroviral Therapy (HAART) on Lean Body Mass
Brief Title: A Study to Evaluate the Effect of Anti-HIV Therapy on Lean Tissue (Muscle) in HIV-Positive Patients
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 892
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-08

CONDITIONS: HIV Infections
Keywords: HIV-1; Muscles; RNA, Viral; Body Composition; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
The purpose of this study is to determine whether HIV-positive patients with extremely low viral loads (level of HIV in the blood) have a greater gain in lean tissue during anti-HIV (antiretroviral) therapy than patients with higher viral loads.

Many HIV-positive patients experience changes in body composition (muscle, fat, etc.) while on antiretroviral therapy. However, any weight gained while taking antiretrovirals is mostly fat. A patient's viral load may affect whether weight gained is a result of increased fat or increased muscle. A large-scale study is needed to closely evaluate the effects of antiretroviral therapy on body composition.

DETAILED DESCRIPTION:
Effective antiretroviral therapy, as measured by a decrease in HIV-1 RNA levels, may sustain or improve important components of body composition, perhaps through a decrease in the underlying pro-inflammatory activity and resting energy expenditure. Moderate weight gain has been reported to be associated with HAART. Meaningful increase in total body weight, however, may need to be comprised of augmentation of lean body mass (primarily muscle), since mortality in HIV and cancer wasting is associated with sizable decreases in lean body mass (LBM) and there is no evidence that increases in fat cell mass are protective. To date, there has not been any large-scale prospective evaluation of the effects of HAART on body composition. Nor has it been determined whether increasing body weight or specific components of body composition (fat or lean body mass) in persons who have lost substantive amounts of weight protects against AIDS-defining complications or prolongs survival.

This is a 48-week, observational study of lean body mass, appetite, functional performance, and systemic markers of inflammation during highly active antiretroviral therapy (HAART) in patients co-enrolled in ACTG antiretroviral studies. Patients are stratified by body mass index (BMI) into 2 cohorts: less than 23 kg/m2 versus greater than or equal to 23 to 28 kg/m2. At selected study visits, times of antiretroviral medication change, and following the diagnosis of an AIDS-defining event, the following are assessed: height (screening visit only), weight, lean body mass, appetite (by questionnaire), functional performance (by questionnaire), and markers of systemic inflammation.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are enrolled in an adult AIDS clinical trial.
* Are HIV-positive.
* Have a viral load of at least 10,000 copies/ml.
* Are expected to live at least 6 months.
* Are at least 18 years old.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Have a history of diabetes requiring medication.
* Have a history of heart disorders.
* Have a fever, diarrhea, nausea, or a condition which makes it difficult to eat within the 14 days prior to study entry.
* Have swelling due to any cause.
* Are pregnant or breast-feeding.
* Are receiving any therapy to increase your appetite or gain weight within 30 days prior to study entry.
* Are receiving any therapy for a severe infection or medical illness within 14 days prior to study entry.
* Are taking certain medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Overall Officials: C Shikuma, Study Chair; D Mildvan, Study Chair; F Sattler, Study Chair
Locations (21):
- United States (20):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ Med Ctr, Stanford, California
  - Howard Univ, Washington D.C., District of Columbia
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Northwestern Univ Med School, Chicago, Illinois
  - Cook County Hosp, Chicago, Illinois
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Beth Israel Med Ctr, New York, New York
  - Chelsea Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Pennsylvania at Philadelphia, Philadelphia, Pennsylvania
  - Univ of Washington, Seattle, Washington
- Univ of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Background] Sattler FR, Schroeder ET, Dube MP, Jaque SV, Martinez C, Blanche PJ, Azen S, Krauss RM. Metabolic effects of nandrolone decanoate and resistance training in men with HIV. Am J Physiol Endocrinol Metab. 2002 Dec;283(6):E1214-22. doi: 10.1152/ajpendo.00189.2002. Epub 2002 Aug 27. PMID 12388173
- [Background] Shikuma CM, Zackin R, Sattler F, Mildvan D, Nyangweso P, Alston B, Evans S, Mulligan K; AIDS Clinical Trial Group 892 Team. Changes in weight and lean body mass during highly active antiretroviral therapy. Clin Infect Dis. 2004 Oct 15;39(8):1223-30. doi: 10.1086/424665. Epub 2004 Sep 27. PMID 15486848